CLINICAL TRIAL: NCT01539304
Title: Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of "CITUS Dry Syrup" in Children With Perennial Allergic Rhinitis: Double Blinded, Randomized, Placebo Controlled, Parallel Designed, Multi-centered, Phase III Study
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of "CITUS Dry Syrup" in Children With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SamA Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CITUS_P3
Record Dates: First submitted 2012-02-06; First posted 2012-02-27 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- CITUS Dry Syrup (Experimental): Pranlukast dry syrup 10%
  Interventions: Drug: CITUS Dry Syrup
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CITUS Dry Syrup — Pranlukast 10% dry syrup, b.i.d.
  Arms: CITUS Dry Syrup
Drug: Placebo — Placebo dry syrup, b.i.d
  Arms: Placebo

SUMMARY:
Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of "CITUS Dry Syrup" in Children With Perennial Allergic Rhinitis: Double Blinded, Randomized, Placebo Controlled, Parallel Designed, Multi-centered, Phase III Study.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged over 24 months and under 15 years.
2. Patients who was diagnosed with perennial allergic rhinitis by ImmunoCAP test.
3. NIS mean total score of 1-week in baseline should be over 4.0.

Exclusion Criteria:

1. Patient who is accompanied by the seriously abnormal symptom in respiratory system, such as pneumonia, cystic fibrosis, viral influenza, tuberculosis, asthma(status praesens).
2. Patient who has cancer, diabetes mellitus, hypertension, CNS disease, and metabolic disease which need medication.
3. Patient who has rhinitis not caused by allergy.
4. Acute or chronic sinusitis.
5. Patient who has medical history of allergy in seasonal pollen during the trial.
6. Patient who has had eyes or nose surgery within 3 months prior to the trial.
7. Patient who has had eye or upper airway infection within 1 week prior to the treatment period.
8. Beginning immunotherapy or dose of change within 1 month prior to the trial.
9. Patient who has clinical history of sensitivity to allergic rhinitis medication.
10. Patient whose heart function is abnormal: including heart failure, abnormal ECG test value that is clinically significant.
11. Patient who has experience to have participated in other clinical trial within 2 months prior to the trial.
12. Patient who has taken contraindicated medications in this study within 1 week(baseline period) prior to the treatment period.
13. For girl who had her first period, result of pregnancy test was positive.

Ages: 24 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in NIS(Nasal Index Score) over the 4-week treatment period | 4 week treatment period (from baseline through the end of week 4)
  Evaluation : from baseline(1-week prior to treatment)over the 4-week treatment(1-week prior to patients' last visit).
  NIS : Sum of 4 individual scores for Nasal congestion, Rhinorrhea, Sneezing, and Nasal itching, each rated by patients daily on a 4-point scale [Score 0(best) to 3(worst)].

SECONDARY OUTCOMES:
Assessing improvement of symptom by physician | from baseline through the end of week 4
Assessing improvement of symptom by patient | from baseline through the end of week 4
Mean change of Individual NIS | from baseline through the end of week 4
Ratio distribution of NIS at end of week 4 | from baseline through the end of week 4
  Percentage of each NIS score.
Cure rate | from baseline through the end of week 4
Cure rate for each symptom | from baseline through the end of week 4
Use of rescue medication | from baseline through the end of week 4
Change of Instantaneous NIS | from baseline through the end of week 4

CONTACTS AND LOCATIONS:
Overall Officials: Young Yull Koh, MD, Principal Investigator — Seoul National University Hospital; Bok Yang Pyun, MD, Principal Investigator — Soonchunhyang University Hospital; Jae Won Oh, MD, Principal Investigator — Hanyang University Guri Hospital; Yeong Ho Na, MD, Principal Investigator — Kyunghee University Medical Center; Soo Jong Hong, MD, Principal Investigator — Asan Medical Center; Hyun Hee Kim, MD, Principal Investigator — The Catholic University of Korea Bucheon St.Mary's Hospital; Dae Hyun Lim, MD, Principal Investigator — Inha University Hospital; Kang Mo Ahn, MD, Principal Investigator — Samsung Medical Center; Myung Hyun Sohn, MD, Principal Investigator — Severance Hospital; Jin Tack Kim, MD, Principal Investigator — The Catholic University of Korea, Uijeongbu ST. Mary's Hospital
Locations (1):
- Seoul National University Hodpital, Seoul, South Korea